CLINICAL TRIAL: NCT03127098
Title: Phase 1b/2 Study of ETBX-011 (Ad5 [E1-, E2b-]-CEA(6D)) Vaccine in Combination With ALT-803 (Super-agonist IL-15) in Subjects Having CEA-Expressing Cancer
Brief Title: QUILT-3.040: ETBX-011 (Ad5 [E1-, E2b-]-CEA(6D)) Vaccine in Combination With ALT-803 (Super-agonist IL-15) in Subjects Having CEA-Expressing Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated before any dose escalation occurred in order to pursue other studies designed to more extensively evaluate the combination of ETBX-011 and N-803 along with other immunotherapy agents.
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.040
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2019-08

CONDITIONS: Thyroid Cancer; Colon Cancer; Ovarian Cancer; Breast Cancer; Lung Cancer; Pancreatic Cancer
Keywords: locally advanced or metastatic; carcinoembryonic antigen (CEA)-expressing; CEA; carcinoembryonic antigen
MeSH Terms: conditions — Thyroid Neoplasms; Colonic Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Presenilin-1; methyl N-acetylsibirosaminide; ALT-803; Interleukin-15

STUDY DESIGN:
Intervention Model Description: ETBX-011 immunization was administered by subcutaneous (SC) injection. ALT-803 will be administered by SC injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ETBX-011 in combination with ALT-803 (Experimental): A combination of agents were administered to subjects in this dose-escalation study
  Interventions: Biological: ETBX-011; Biological: ALT-803

INTERVENTIONS:
Biological: ETBX-011 — ETBX-011 immunization was administered by subcutaneous (SC) injection.
  Other Names: Ad5 [E1-, E2b-]-CEA(6D)
Biological: ALT-803 — ALT-803 was administered by SC injection.
  Other Names: Super-agonist IL-15; IL-15

SUMMARY:
This is a phase 1b/2 study to evaluate the safety, tolerability, and efficacy of ETBX-011 vaccine used in combination with ALT-803 in subjects with locally advanced or metastatic CEA-expressing cancers whose tumor has recurred after standard-of-care treatment.

DETAILED DESCRIPTION:
The trial will consist of a phase 1b study with ETBX-011 as a fixed dose with a dose escalation of ALT-803 unless de-escalation is required. The proposed phase 2 expansion study will give additional safety data for the MTD as well as preliminary efficacy data. Subjects will receive treatments unless they experience progressive disease, dose-limiting toxicities (DLT), withdraw consent, or if the investigator determines it is no longer in their best medical interest to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 21 years.
2. Subjects with a histologically confirmed diagnosis of locally advanced or metastatic malignancy who were previously treated with at least one method of standard therapy known to have a possible survival benefit or refused such therapy.
3. The tumor must express CEA or must be known to be universally CEA positive (ie, colon and rectal cancer).
4. Must have a recent FFPE tumor biopsy specimen.
5. Subjects who have received prior CEA-targeted immunotherapy (eg, vaccine or antibody) are eligible for this trial if this treatment was discontinued at least 3 months prior to enrollment.
6. Resolution of all toxic side effects of prior chemotherapy, radiotherapy, or surgical procedures to NCI CTCAE grade ≤ 1.
7. Ability to understand and provide signed informed consent that fulfills Institutional Review Board (IRB)'s guidelines.
8. ECOG performance status of 0 or 1.
9. Subjects who are taking medications that do not have a known history of immunosuppression are eligible for this trial.
10. Adequate hematologic function at screening, as follows:
11. WBC count ≥ 3000/microliter.
12. Hemoglobin ≥ 9 g/dL (may not transfuse or use erythropoietin to achieve this level).
13. Platelets ≥ 75,000/microliter.
14. Prothrombin (PT)-international normalized ratio (INR) < 1.5.
15. Partial thromboplastin time (PTT) < 1.5 × upper limit of normal (ULN).
16. Adequate renal and hepatic function at screening, as follows:
17. Serum creatinine < 2.0 mg/dL.
18. Bilirubin < 1.5 mg/dL (except for Gilbert's syndrome which will allow bilirubin ≤ 2.0 mg/dL).
19. Alanine aminotransferase (ALT) ≤ 2.5 × ULN.
20. Aspartate aminotransferase (AST) ≤ 2.5 × ULN.
21. Female subjects of childbearing potential and women < 12 months since the onset of menopause must agree to use acceptable contraceptive methods for the duration of the study and for 7 months following the last injection of study medication. Male subjects must be surgically sterile or must agree to use a condom and acceptable contraceptive method with their partner.
22. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.

Exclusion Criteria:

1. Participation in an investigational drug or device study within 30 days of screening for this study.
2. Pregnant and nursing women.
3. Subjects with ongoing everolimus or other cancer therapy that interferes with the induction of immune responses.
4. Subjects with concurrent cytotoxic chemotherapy or radiation therapy. There must be at least one (1) month between any other prior chemotherapy (or radiotherapy) and study treatment. Any prior CEA-targeted immunotherapy (vaccine) must have been discontinued at least 3 months before initiation of study treatment. Subjects must have recovered from all acute toxicities from prior treatment prior to screening for this study.
5. Active brain or central nervous system metastasis, seizures requiring anticonvulsant treatment, cerebrovascular accident (< 6 months), or transient ischemic attack.
6. Subjects with a history of autoimmune disease (active or past), such as but not restricted to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Autoimmune-related thyroid disease and vitiligo are permitted.
7. Subjects with serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, or other illness considered by the Investigator as high risk for investigational drug treatment.
8. Subjects with a history of heart disease, such as congestive heart failure (class II, III, or IV defined by the New York Heart Association functional classification), history of unstable or poorly controlled angina, or history (< 1 year) of ventricular arrhythmia.
9. Subjects with a medical or psychological impediment that would impair the ability of the subject to receive therapy per protocol or impact ability to comply with the protocol or protocol-required visits and procedures.
10. History of malignancy except for the following: adequately treated non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other carcinoma that has been in complete remission without treatment for more than 5 years.
11. Presence of a known active acute or chronic infection, including human immunodeficiency virus (HIV, as determined by enzyme-linked immunosorbent assay [ELISA] and confirmed by western blot) and hepatitis B and hepatitis C virus (HBV/HCV, as determined by HBsAg and hepatitis C serology).
12. Subjects on systemic intravenous or oral steroid therapy (or other immunosuppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Subjects must have had at least 6 weeks of discontinuation of any steroid therapy (except that used as premedication for chemotherapy or contrast-enhanced studies) prior to enrollment.
13. Subjects with known allergy or hypersensitivity to any component of the investigational product will be excluded.
14. Subjects with acute or chronic skin disorders that will interfere with injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
15. Subjects vaccinated with a live (attenuated) vaccine (e.g., FluMist®) or a killed (inactivated)/subunit vaccine (e.g., PNEUMOVAX®, Fluzone®) within 28 days or 14 days, respectively, of the first planned dose of ETBX-011 or ALT 803.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology Associates, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the first dose level, N-803 10 μg/kg/dose + ETBX-011 (5 × 10^11 VP/dose), was administered due to study termination. No additional escalations or the expansion phase (Phase 2) occurred.
  No patients had a response, therefore, Duration of Response could not be summarized.
  Only 2 out of 3 enrolled patients had a response assessment data, therefore, Progression Free Survival and Overall Survival analyses will not provide a meaningful result.
Period: Overall Study
Arm/Group | ETBX-011 in Combination With ALT-803
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ETBX-011 in Combination With ALT-803
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Subjects with previously treated locally advanced or metastatic CEA-expressing cancer [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ETBX-011 in Combination With ALT-803
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Duration of Response
Description: The duration of overall response was measured from the time measurement criteria are met for CR or PR (whichever was first recorded) until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started).
Time Frame: Up to 11 weeks
Population: No objective responses were observed.
Arm/Group | ETBX-011 in Combination With ALT-803
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurred first. Subjects who did not have disease progression or did not die at the end of follow up were to be censored at the last known date the subject was progression free.
Time Frame: Up to 11 weeks
Population: No objective responses were observed.
Measure: Count of Participants; unit: Participants
Arm/Group | ETBX-011 in Combination With ALT-803
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Overall Survival
Description: OS was evaluated by dose cohort and overall using the Kaplan-Meier method. OS was defined as the time from the date of first treatment to the date of death from any cause. Subjects who were alive at the end of follow up were to be censored at the last known date alive.
Time Frame: Up to 6 months
Population: No objective responses were observed.
Measure: Number; unit: Months
Arm/Group | ETBX-011 in Combination With ALT-803
Number analyzed (Participants) | 3
Months | NA — insufficient number of participants with event

ADVERSE EVENTS:
Time Frame: Non-serious AEs were to be followed for 30 days after subject's last dose of ETBX-011+ALT-803, up to 13 weeks . Non-serious grade 3/4 AEs were to be followed until resolution or stabilization, up to 13 weeks. All SAEs that did not resolve upon discontinuation of the subject's participation in the study were to be followed until recovered, recovered w/ sequelae, lost to follow-up, otherwise, up to 13 weeks. All-Cause Mortality was assessed through study completion, up to 6 months.
Arm/Group | ETBX-011 in Combination With ALT-803
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETBX-011 in Combination With ALT-803 (N=3)
Lymph node pain (Blood and lymphatic system disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 2
Influenza like illness (General disorders) | 2
Injection site erythema (General disorders) | 3
Injection site oedema (General disorders) | 3
Injection site pain (General disorders) | 3
Injection site pruritus (General disorders) | 3
Pyrexia (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03127098/Prot_SAP_000.pdf